CLINICAL TRIAL: NCT02784873
Title: High Intensity Interval Training (HIIT) Versus Moderate Intensity Steady State Training (MISS) in UK Cardiac Rehabilitation Programmes: a Multi-centre Randomised Controlled Trial and Economic Evaluation
Brief Title: High Intensity Interval Training in UK Cardiac Rehabilitation Programmes
Acronym: HIIT-or-MISS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: Cardiff Metropolitan University (Other); City Health Care Partnership CIC (Hull) (Unknown); University of Hull (Other); Aneurin Bevan University Health Board (Other); Wake Forest University Health Sciences (Other); Bangor University (Other); University of Warwick (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GM164715
Record Dates: First submitted 2016-03-24; First posted 2016-05-27 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Coronary Disease
Keywords: High intensity interval training; Coronary heart disease; Exercise training; Cardiac rehabilitation; Interval training
MeSH Terms: conditions — Coronary Disease | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Usual care cardiac rehabilitation with exercise training as per current guidelines
  Warm up: 15 mins, < 40% heart rate reserve (HRR) Cardiovascular component: progress towards 20 - 40 mins continuous cardiovascular exercise at 40-70% HRR.
  Muscular strength and endurance programme. Cool down: 10 mins, < 40% HRR. Initial duration based on participant's previous and current physical activity (PA) levels and cardiopulmonary exercise test (CPEX) performance.
  Duration and workload of cardiovascular component adjusted, as tolerated, within the above parameters, in response to exercising heart rate (HR), participant reported rating of perceived exertion (RPE) and symptoms.
- High intensity interval training (Experimental): High intensity interval training within a standard cardiac rehabilitation programme.
  Warm up: 15 mins total, 10 mins <40-70% HRR, 5 mins <70% HRR. Cardiovascular component: exercise bike interval training: 10 x high @ 85-90% peak power output (PPO) from CPEX, 10 x low @ 20-25% PPO (exercise intensity will not to be prescribed from gas exchange data i.e. %VO2 peak). Change in intensity from low to high achieved by altering cadence (rpm).
  Muscular strength and endurance programme. Cool down: 10 mins, <40% HRR. Duration of intervals and total programme duration increased in a standardised fashion.
  Workload increased bi-weekly in response to participant reported RPE (only after the full 10 x 1 protocol has been achieved). If RPE < 17 then workload will be increased.
  Interventions: Other: High intensity interval training

INTERVENTIONS:
Other: High intensity interval training — High intensity interval training within a standard cardiac rehabilitation programme
  Arms: High intensity interval training

SUMMARY:
The purpose of the trial is to compare the effects of high intensity interval training (HIIT) with usual care - moderate intensity steady state training (MISS) - in UK cardiac rehabilitation (CR) programmes.

DETAILED DESCRIPTION:
Current cardiac rehabilitation (CR) guidelines recommend moderate intensity, steady state exercise training (MISS). However, this guideline predates significant advances in interventional and medical treatment for coronary heart disease (CHD) and may not, therefore, be the most effective strategy for the 'modern' patient with CHD. Recent research has indicated that greater benefit may be attained by participating in high intensity interval training (HIIT) which involves repeated short bursts of harder exercise interspersed with short recovery periods. Studies suggest that this can be performed without any compromise in exercise adherence or patient safety. The benefit of this approach in 'real world' CR programmes in the UK cannot be confirmed, as studies have been predominantly conducted in the laboratory and exclusively outside the UK.

In patients attending CR programmes in the UK, the investigators hypothesise that HIIT will improve VO2 peak to a greater extent than MISS. The investigators also hypothesise that HIIT will: 1) be more palatable than MISS and demonstrate greater patient compliance and adherence; 2) improve cardiovascular health to a greater extent than MISS; 3) improve HR-QoL to a greater extent than MISS; 4) lead to more positive motivation and attitudes to exercise than MISS; 5) increase short and medium-term participation in lifestyle physical activity to a greater extent than MISS; 6) be a cost effective alternative to MISS; 7) be as safe as MISS.

The HIIT or MISS study is a pragmatic single-blind, multi-centre, longitudinal, randomised controlled trial. Participants will be randomly allocated to 8 weeks of HIIT or MISS (usual care). Outcomes will be assessed at baseline, 8 weeks and 12 months by assessors blinded to group allocation. Study interventions will be delivered by clinical (not research) staff.

ELIGIBILITY:
General inclusion criteria:

1. Successfully revascularised following percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)
2. Angiographically documented non-obstructive coronary artery disease (CAD)
3. Left ventricular ejection fraction (LVEF) > 40%
4. Clinically stable (symptoms and medication) for > 2 weeks 5.18 - 75 yrs of age

General exclusion criteria:

1. Symptoms of ischemia
2. Significant left main stem stenosis
3. NYHA class III-IV symptoms
4. Compromising cardiac ventricular arrhythmia
5. Significant valvular heart disease
6. Inability to comply with guidelines for participation in exercise testing and training
7. Significant limiting comorbidities that would prevent full participation

Additional exclusion criteria:

Further to the analysis of cardiopulmonary exercise test and echocardiography at baseline, and prior to randomisation, patients will be prevented from continuing their involvement in the study if there is indication of:

1. Exercise induced ischemia or significant hemodynamic compromise
2. LVEF < 40%
3. Clinical instability in accordance with CR guidelines
4. Inability to comply with guidelines for participation in exercise testing and training

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Change in peak oxygen uptake (VO2 peak) | Baseline, 8 weeks and 12 months
  Cardiopulmonary exercise test

SECONDARY OUTCOMES:
Compliance and adherence | Every exercise session (8 week exercise programme duration)
  Compliance and adherence will be determined by recording the number of training sessions attended and successfully completed in accordance with the exercise protocol. Drop-out from the programme will also be documented for both study groups in addition to reason for drop-out, where provided voluntarily by participants.
Psychological factors associated with compliance and adherence (1) | Baseline, 8 weeks
  Quantitative psychology - questionnaires: 1) the Multidimensional Self-Efficacy for Exercise Scale (MSES)
Psychological factors associated with compliance and adherence (2) | Baseline, 8 weeks
  Quantitative psychology - questionnaires: 2) the Behavioural Regulation in Exercise Questionnaire-2 (BREQ-2)
Psychological factors associated with compliance and adherence (3) | Baseline, 8 weeks
  Quantitative psychology - questionnaires: 3) the Psychological Need Satisfaction in Exercise Scale (PNSES)
Psychological factors associated with compliance and adherence (4) | Baseline, 8 weeks
  Quantitative psychology - questionnaires: 4) Courneya and Bobick's 7-point bipolar adjectival rating scale;
HR-QOL | Baseline, 8 weeks and 12 months
  Questionnaire - EQ-5D-5L
Service and resource use | Baseline, 8 weeks and 12 months
  Questionnaire - client service receipt inventory (CSRI)
Lifestyle physical activity | Baseline, 8 weeks and 12 months
  Physical activity monitor (worn for 1 week) - total energy expenditure
Metabolic reserve | Baseline, 8 weeks and 12 months
  Cardiopulmonary exercise test - ventilatory threshold (VT)
Ventilatory efficiency | Baseline, 8 weeks and 12 months
  Cardiopulmonary exercise test - slope of ratio of ventilation to carbon dioxide (VE/VC02 slope)
Cardiac remodelling | Baseline, 8 weeks and 12 months
  Echocardiography - left ventricular volumes
Arterial remodelling | Baseline, 8 weeks and 12 months
  Arterial oscillometry - pulse wave velocity
Cardiovascular health | Baseline, 8 weeks and 12 months
  CHD risk factor assessment
Palatability | 8 weeks
  Qualitative psychology - thematic analysis of semi structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Karianne Backx, PhD, Principal Investigator — Cardiff Metropolitan University; Simon Nichols, PhD, Principal Investigator — University of Hull
Locations (1):
- University Hospital, Coventry, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] West RR, Jones DA, Henderson AH. Rehabilitation after myocardial infarction trial (RAMIT): multi-centre randomised controlled trial of comprehensive cardiac rehabilitation in patients following acute myocardial infarction. Heart. 2012 Apr;98(8):637-44. doi: 10.1136/heartjnl-2011-300302. Epub 2011 Dec 22. PMID 22194152
- [Background] Liou K, Ho S, Fildes J, Ooi SY. High Intensity Interval versus Moderate Intensity Continuous Training in Patients with Coronary Artery Disease: A Meta-analysis of Physiological and Clinical Parameters. Heart Lung Circ. 2016 Feb;25(2):166-74. doi: 10.1016/j.hlc.2015.06.828. Epub 2015 Jul 22. PMID 26375499
- [Background] Elliott AD, Rajopadhyaya K, Bentley DJ, Beltrame JF, Aromataris EC. Interval training versus continuous exercise in patients with coronary artery disease: a meta-analysis. Heart Lung Circ. 2015 Feb;24(2):149-57. doi: 10.1016/j.hlc.2014.09.001. Epub 2014 Sep 16. PMID 25306500
- [Background] Rognmo O, Moholdt T, Bakken H, Hole T, Molstad P, Myhr NE, Grimsmo J, Wisloff U. Cardiovascular risk of high- versus moderate-intensity aerobic exercise in coronary heart disease patients. Circulation. 2012 Sep 18;126(12):1436-40. doi: 10.1161/CIRCULATIONAHA.112.123117. Epub 2012 Aug 9. PMID 22879367
- [Derived] Ingle L, Powell R, Begg B, Birkett ST, Nichols S, Ennis S, Banerjee P, Shave R, McGregor G. Effects of Exercise Training Response on Quality of Life and Cardiovascular Risk Factor Profiles in People With Coronary Artery Disease: Insights From the HIIT or MISS UK Trial. Arch Phys Med Rehabil. 2024 Aug;105(8):1464-1470. doi: 10.1016/j.apmr.2024.03.002. Epub 2024 Mar 16. PMID 38493909
- [Derived] Albustami M, Hartfiel N, Charles JM, Powell R, Begg B, Birkett ST, Nichols S, Ennis S, Hee SW, Banerjee P, Ingle L, Shave R, McGregor G, Edwards RT. Cost-effectiveness of High-Intensity Interval Training (HIIT) vs Moderate Intensity Steady-State (MISS) Training in UK Cardiac Rehabilitation. Arch Phys Med Rehabil. 2024 Apr;105(4):639-646. doi: 10.1016/j.apmr.2023.09.005. Epub 2023 Sep 18. PMID 37730193
- [Derived] McGregor G, Powell R, Begg B, Birkett ST, Nichols S, Ennis S, McGuire S, Prosser J, Fiassam O, Hee SW, Hamborg T, Banerjee P, Hartfiel N, Charles JM, Edwards RT, Drane A, Ali D, Osman F, He H, Lachlan T, Haykowsky MJ, Ingle L, Shave R. High-intensity interval training in cardiac rehabilitation: a multi-centre randomized controlled trial. Eur J Prev Cardiol. 2023 Jul 12;30(9):745-755. doi: 10.1093/eurjpc/zwad039. PMID 36753063
- [Derived] McGregor G, Nichols S, Hamborg T, Bryning L, Tudor-Edwards R, Markland D, Mercer J, Birkett S, Ennis S, Powell R, Begg B, Haykowsky MJ, Banerjee P, Ingle L, Shave R, Backx K. High-intensity interval training versus moderate-intensity steady-state training in UK cardiac rehabilitation programmes (HIIT or MISS UK): study protocol for a multicentre randomised controlled trial and economic evaluation. BMJ Open. 2016 Nov 16;6(11):e012843. doi: 10.1136/bmjopen-2016-012843. PMID 27852718